CLINICAL TRIAL: NCT03498586
Title: Half-normal Saline vs Normal Saline for Irrigation of Open-irrigated Radiofrequency Catheters in Atrial Fibrillation Ablation
Brief Title: Half-normal Saline in Atrial Fibrillation Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Responsible Party: Principal Investigator, Andrea Natale, Executive Medical Director, Texas Cardiac Arrhythmia Research Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TCAI_HNS_AF
Record Dates: First submitted 2018-04-04; First posted 2018-04-13 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Half-normal saline (Experimental)
  Interventions: Drug: Half-normal saline
- Normal saline (Active Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Half-normal saline — Use of half-normal saline as an irrigant for open-irrigated ablation catheters
  Arms: Half-normal saline
Drug: Normal saline — Use of normal saline as an irrigant for open-irrigated ablation catheters
  Arms: Normal saline

SUMMARY:
The study evaluates the use of half-normal saline as an irrigant for open-irrigated catheters during atrial fibrillation ablation. By increasing the efficacy of radiofrequency energy-mediated lesion formation, half-normal saline has the potential to reduce procedural times and improved acute and long-term outcomes.

ELIGIBILITY:
Inclusion criteria

* male or female between 18 and 75 years of age at the time of enrollment
* undergoing first-time radiofrequency ablation for atrial fibrillation
* written informed consent obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study

Exclusion criteria

* robotic-guided atrial fibrillation ablation
* baseline hyponatremia (serum sodium level < 135 mEq/L)
* pregnant, breastfeeding, or unwilling to practice birth control during participation in the study
* presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2020-05-02 (Actual)

PRIMARY OUTCOMES:
total radiofrequency ablation time, and total procedure time | intraprocedural
acute pulmonary veins, and left atrial appendage (if applicable) reconnection | intraprocedural
freedom from atrial tachycardia/atrial fibrillation > 30 seconds without antiarrhythmic drugs | 1 year

SECONDARY OUTCOMES:
freedom from atrial tachycardia/atrial fibrillation > 30 seconds with or without antiarrhythmic drugs | 1 year
long-term pulmonary veins, left atrial appendage (if applicable), and coronary sinus (if applicable) reconnection | in case of a repeat procedure performed during the study follow-up (an average of 1 year)

OTHER OUTCOMES:
procedure-related complications | periprocedural (at the time of the procedure and up to 1 month)
  pericardial effusion due to cardiac perforation or pericarditis, transient ischemic attack/stroke, systemic embolism, phrenic nerve injury, pulmonary vein stenosis, atrio-esophageal fistula, death
hyponatremia | periprocedural (at the time of the procedure and up to 1 month)
  serum sodium level < 135 mEq/L

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, MD, Principal Investigator — Texas Cardiac Arrhythmia Institute, St. David's Medical Center
Locations (2):
- Texas Cardiac Arrhythmia Institute, St. David's Medical Center, Austin, Texas, United States
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada